CLINICAL TRIAL: NCT02137785
Title: A Phase 3 Study of Photodynamic Therapy With Levulan Kerastick Topical Solution + Blue Light Versus Topical Solution Vehicle + Blue Light for the Treatment of Actinic Keratoses on the Upper Extremities
Brief Title: Safety and Efficacy Study of Photodynamic Therapy With Levulan Kerastick + Blue Light for Actinic Keratoses on the Upper Extremities
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: DUSA Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP0108
Record Dates: First submitted 2014-05-07; First posted 2014-05-14 (Estimated); Results first posted 2015-09-16 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-08

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Aminolevulinic Acid; Solutions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALA (Experimental)
  Interventions: Drug: Aminolevulinic Acid (ALA); Device: Blue Light Photodynamic Therapy Illuminator (BLU-U)
- Vehicle (Placebo Comparator)
  Interventions: Drug: Topical Solution Vehicle; Device: Blue Light Photodynamic Therapy Illuminator (BLU-U)

INTERVENTIONS:
Drug: Aminolevulinic Acid (ALA) — 20% ALA applied to upper extremities for 3 hours prior to 10 J/cm2 blue light
  Other Names: Levulan Kerastick
  Arms: ALA
Drug: Topical Solution Vehicle — Levulan Kerastick containing vehicle ingredients only. Vehicle solution applied to upper extremities 3 hours prior to 10 J/cm2 blue light
  Arms: Vehicle
Device: Blue Light Photodynamic Therapy Illuminator (BLU-U) — 10 J/cm2 blue light delivered at 10mW/cm2

SUMMARY:
The purpose of this study is to determine if Levulan Photodynamic Therapy (PDT) is safe and effective in the treatment of actinic keratoses on the upper arms and hands

ELIGIBILITY:
Inclusion Criteria:

* Four to fifteen Grade 1/2 actinic keratosis lesions (AKs) on one upper extremity

Exclusion Criteria:

* Pregnancy
* grade 3 and/or atypical >1cm AKs within Treatment Area
* history of cutaneous photosensitization, porphyria, hypersensitivity to porphyrins or photodermatosis
* lesions suspicious for skin cancer (skin cancer not ruled out by biopsy) or untreated skin cancers within the Treatment Area
* skin pathology or condition which could interfere with the evaluation of the test product or requires the use of interfering topical or systemic therapy
* Subject is immunosuppressed
* unsuccessful outcome from previous ALA-PDT therapy
* currently enrolled in an investigational drug or device study
* has received an investigational drug or been treated with an investigational device within 30 days prior to the initiation of treatment
* known sensitivity to one or more of the vehicle components (ethyl alcohol, isopropyl alcohol, laureth 4, polyethylene glycol)
* use of the following topical preparations on the extremity to be treated:

  * Keratolytics including urea (greater than 5%), alpha hydroxyacids [e.g.glycolic acid, lactic acid, etc. greater than 5%], salicylic acid (greater than 2%) within 2 days of initiation of treatment.
  * Cryotherapy within 2 weeks of initiation of treatment
  * Retinoids, including tazarotene, adapalene, tretinoin, within 4 weeks of initiation of treatment.
  * Microdermabrasion, laser ablative treatments, ALA-PDT, chemical peels, 5-FU, diclofenac, ingenol mebutate, imiquimod or other topical treatments for AK within 8 weeks of initiation of treatment.
* use of systemic retinoid therapy within 6 months of initiation of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2014-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Marcus, MD, PhD, Study Director — DUSA Pharmaceuticals, Inc.
Locations (13):
- United States (13):
  - Center For Dermatology Clinical Research, Inc., Fremont, California
  - UCSD Dermatology, San Diego, California
  - Center for Clinical and Cosmetic Research, Aventura, Florida
  - MOORE Clinical Research, Inc, Brandon, Florida
  - Spencer Clinical Services, St. Petersburg, Florida
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - Shideler Clinical Research Center, Carmel, Indiana
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Oregon Dermatology and Research Center, Portland, Oregon
  - J&S Studies, Inc, College Station, Texas
  - Suzanne Bruce and Associates, P.A.,The Center for Skin Research, Houston, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia

REFERENCES:
- [Derived] Piacquadio D, Berman B, Siegel DM, Bhatia N, Brocato J, Squittieri N, Pariser DM. Treatment Satisfaction and Acceptability of 20% Aminolevulinic Acid Photodynamic Therapy for the Treatment of Actinic Keratoses of the Face, Scalp, and Upper Extremities. J Clin Aesthet Dermatol. 2023 Dec;16(12):46-51. PMID 38125671

RESULTS

PARTICIPANT FLOW:
Groups:
- ALA-PDT: Aminolevulinic Acid (ALA): 20% ALA applied to upper extremities for 3 hours prior to 10 J/cm2 blue light
  BLU-U Blue Light Photodynamic Therapy Illuminator: 10 J/cm2 blue light delivered at 10mW/cm2
- Vehicle: Topical Solution Vehicle: Levulan Kerastick containing vehicle ingredients only. Vehicle solution applied to upper extremities 3 hours prior to 10 J/cm2 blue light
  BLU-U Blue Light Photodynamic Therapy Illuminator: 10 J/cm2 blue light delivered at 10mW/cm2
Period: Overall Study
Arm/Group | ALA-PDT | Vehicle
Started | 135 | 134
Completed | 132 | 130
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 4
Not completed — subject moved out of state | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT
Groups:
- Total: Total of all reporting groups
Arm/Group | ALA-PDT | Vehicle | Total
Number analyzed (Participants) | 135 | 134 | 269
Age, Continuous [Mean (Full Range); unit: years] | 67.6 [45 to 90] | 67.6 [47 to 87] | 67.6 [45 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 38 | 81
  Male | 92 | 96 | 188
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 135 | 131 | 266
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 135 | 134 | 269
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Skin Type [Number; unit: participants] — Fitzpatrick Skin Type I - Always burns easily; never tans (sensitive) II - Always burns easily; tans minimally (sensitive) III - Burns moderately; tans gradually (light brown) (normal) IV - Burns minimally, always tans well (moderate brown) (normal) V - Rarely burns; tans profusely (dark brown) (insensitive) VI - Never burns; deeply pigmented (insensitive)
  participants
    Type I | 17 | 16 | 33
    Type II | 67 | 73 | 140
    Type III | 37 | 32 | 69
    Type IV | 14 | 13 | 27
    Type V | 0 | 0 | 0
    Type VI | 0 | 0 | 0
Total Number AK Lesions (Grade 1/2) [Mean (Standard Deviation); unit: lesions per subject] | 8.5 (3.6) | 8.6 (3.4) | 8.5 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Complete Clearance Rate
Description: proportion of subjects in each treatment group with a count of zero lesions in the Treatment Area
Time Frame: Week 12
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants | 42 | 17
Statistical Analysis 1: Comparison: ALA-PDT vs Vehicle; A hierarchical procedure was used to control the level of significance. If the primary analysis was sig (p≤0.05), then AKCR at Week 12 were to be compared. If this analysis was significant, then the AKCR at Week 8 were to be compared. If this analysis was significant, then the CCR at Week 8 was to be compared; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel — Analysis uses observed data only. Missing data was not imputed except for subjects with missing CCR are classified as not having a CCR (ie non-responder); CMH test stratified by analysis center

2. Secondary Outcome: AK Clearance Rate
Description: {1 - [(number of AK lesions at follow-up)/(number of AK lesions at Baseline)]} x 100
Time Frame: Baseline and Week 12
Population: ITT using observed data only
Measure: Mean (Standard Deviation); unit: percentage of baseline lesions cleared
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 132 | 130
percentage of baseline lesions cleared | 69.1 (37.4) | 29.9 (51.5)
Statistical Analysis 1: Comparison: ALA-PDT vs Vehicle; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; linear mixed model with fixed effects for treatment group, time point, and treatment group by time point interaction

3. Secondary Outcome: AK Clearance Rate
Description: {1 - [(number of AK lesions at follow-up)/(number of AK lesions at Baseline)]} x 100
Time Frame: Baseline and Week 8
Population: ITT using observed data only
Measure: Mean (Standard Deviation); unit: percentage of baseline lesions cleared
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 133 | 129
percentage of baseline lesions cleared | 53.4 (45.0) | 26.3 (44.3)
Statistical Analysis 1: Comparison: ALA-PDT vs Vehicle; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; linear mixed model with fixed effects for treatment group, time point, and treatment group by time point interaction

4. Secondary Outcome: Complete Clearance Rate
Description: proportion of subjects in each treatment group with a count of zero lesions in the Treatment Area
Time Frame: Week 8
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants | 35 | 12
Statistical Analysis 1: Comparison: ALA-PDT vs Vehicle; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; CMH test stratified by analysis center

5. Secondary Outcome: Subject Satisfaction Score
Description: Subject satisfaction score
  1. = Excellent (very satisfied)
  2. = Good (moderately satisfied)
  3. = Fair (slightly satisfied)
  4. = Poor (not satisfied at all)
Time Frame: Week 12
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 134 | 131
participants
  Very Satisfied | 71 | 29
  Moderately Satisfied | 47 | 26
  Slightly Satisfied | 12 | 28
  Not Satisfied | 4 | 48

6. Other Pre Specified Outcome: Hyperpigmentation
Description: HYPERPIGMENTATION SCALE Grade 0 = No hyperpigmentation Grade 1 = Light hyperpigmentation involving small areas Grade 2 = Moderate hyperpigmentation involving small areas; light hyperpigmentation involving moderate areas Grade 3 = Moderate hyperpigmentation involving moderate sized areas; light hyperpigmentation involving large areas; small areas of marked hyperpigmentation Grade 4 = Marked hyperpigmentation involving moderate or large sized areas
Time Frame: Baseline
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants
  Grade 0 (none) | 46 | 53
  Grade 1 (light) | 51 | 34
  Grade 2 (moderate - small) | 27 | 35
  Grade 3 (moderate - moderate) | 10 | 10
  Grade 4 (marked) | 1 | 2

7. Other Pre Specified Outcome: Hyperpigmentation
Description: as for outcome 6
Time Frame: 24-48 hours after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants
  Grade 0 (none) | 46 | 58
  Grade 1 (light) | 49 | 34
  Grade 2 (moderate - small) | 28 | 30
  Grade 3 (moderate - moderate) | 11 | 10
  Grade 4 (marked) | 1 | 2

8. Other Pre Specified Outcome: Hyperpigmentation
Description: as for outcome 6
Time Frame: 2 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants
  Grade 0 (none) | 45 | 58
  Grade 1 (light) | 46 | 35
  Grade 2 (moderate - small) | 33 | 30
  Grade 3 (moderate - moderate) | 10 | 9
  Grade 4 (marked) | 1 | 2

9. Other Pre Specified Outcome: Hyperpigmentation
Description: as for outcome 6
Time Frame: 4 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 132
participants
  Grade 0 (none) | 51 | 56
  Grade 1 (light) | 44 | 37
  Grade 2 (moderate - small) | 30 | 28
  Grade 3 (moderate - moderate) | 9 | 9
  Grade 4 (marked) | 1 | 2

10. Other Pre Specified Outcome: Hyperpigmentation
Description: as for outcome 6
Time Frame: 8 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 132 | 129
participants
  Grade 0 (none) | 51 | 53
  Grade 1 (light) | 44 | 37
  Grade 2 (moderate - small) | 27 | 27
  Grade 3 (moderate - moderate) | 9 | 10
  Grade 4 (marked) | 1 | 2

11. Other Pre Specified Outcome: Hyperpigmentation
Description: as for outcome 6
Time Frame: 12 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 132 | 130
participants
  Grade 0 (none) | 52 | 49
  Grade 1 (light) | 42 | 43
  Grade 2 (moderate - small) | 29 | 26
  Grade 3 (moderate - moderate) | 8 | 10
  Grade 4 (marked) | 1 | 2

12. Other Pre Specified Outcome: Hypopigmentation
Description: HYPOPIGMENTATION SCALE Grade 0 = No hypopigmentation Grade 1 = Light hypopigmentation involving small areas Grade 2 = Moderate hypopigmentation involving small areas; light hypopigmentation involving moderate areas Grade 3 = Moderate hypopigmentation involving moderate sized areas; light hypopigmentation involving large areas; small areas of marked hypopigmentation Grade 4 = Marked hypopigmentation involving moderate or large sized areas
Time Frame: Baseline
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants
  Grade 0 (none) | 75 | 64
  Grade 1 (light) | 40 | 47
  Grade 2 (moderate - small) | 16 | 17
  Grade 3 (moderate - moderate) | 4 | 4
  Grade 4 (marked) | 0 | 2

13. Other Pre Specified Outcome: Hypopigmentation
Description: as for outcome 12
Time Frame: 24-48 hours after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants
  Grade 0 (none) | 76 | 68
  Grade 1 (light) | 42 | 46
  Grade 2 (moderate - small) | 12 | 14
  Grade 3 (moderate - moderate) | 5 | 4
  Grade 4 (marked) | 0 | 2

14. Other Pre Specified Outcome: Hypopigmentation
Description: as for outcome 12
Time Frame: 2 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants
  Grade 0 (none) | 74 | 67
  Grade 1 (light) | 44 | 47
  Grade 2 (moderate - small) | 13 | 14
  Grade 3 (moderate - moderate) | 4 | 4
  Grade 4 (marked) | 0 | 2

15. Other Pre Specified Outcome: Hypopigmentation
Description: as for outcome 12
Time Frame: 4 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 132
participants
  Grade 0 (none) | 76 | 65
  Grade 1 (light) | 42 | 47
  Grade 2 (moderate - small) | 13 | 14
  Grade 3 (moderate - moderate) | 4 | 4
  Grade 4 (marked) | 0 | 2

16. Other Pre Specified Outcome: Hypopigmentation
Description: as for outcome 12
Time Frame: 8 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 132 | 129
participants
  Grade 0 (none) | 75 | 63
  Grade 1 (light) | 39 | 45
  Grade 2 (moderate - small) | 15 | 15
  Grade 3 (moderate - moderate) | 3 | 4
  Grade 4 (marked) | 0 | 2

17. Other Pre Specified Outcome: Hypopigmentation
Description: as for outcome 12
Time Frame: 12 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 132 | 130
participants
  Grade 0 (none) | 73 | 66
  Grade 1 (light) | 40 | 45
  Grade 2 (moderate - small) | 16 | 14
  Grade 3 (moderate - moderate) | 3 | 3
  Grade 4 (marked) | 0 | 2

18. Other Pre Specified Outcome: Erythema
Description: Erythema Scale - Grade 0 = None Grade 1 = Minimal - barely perceptible erythema Grade 2 = Mild - predominantly minimal erythema (pink) in the treated area with or without a few isolated areas of more intense erythema Grade 3 = Moderate - predominantly moderate erythema (red) in the treated area with or without a few isolated areas of intense erythema (bright red) Grade 4 = Severe - predominantly intense erythema (bright red) in the treated area with or without a few isolated areas of very intense (fiery red) erythema
Time Frame: Baseline
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants
  Grade 0 (none) | 73 | 73
  Grade 1 (minimal) | 38 | 39
  Grade 2 (mild) | 21 | 19
  Grade 3 (moderate) | 3 | 3
  Grade 4 (severe) | 0 | 0

19. Other Pre Specified Outcome: Erythema
Description: as for outcome 18
Time Frame: 5 minutes after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants
  Grade 0 (none) | 12 | 57
  Grade 1 (light) | 26 | 41
  Grade 2 (mild) | 43 | 27
  Grade 3 (moderate) | 52 | 9
  Grade 4 (severe) | 2 | 0

20. Other Pre Specified Outcome: Erythema
Description: as for outcome 18
Time Frame: 24-48 hours after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants
  Grade 0 (none) | 2 | 64
  Grade 1 (minimal) | 16 | 43
  Grade 2 (mild) | 48 | 23
  Grade 3 (moderate) | 66 | 4
  Grade 4 (severe) | 3 | 0

21. Other Pre Specified Outcome: Erythema
Description: as for outcome 18
Time Frame: 2 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants
  Grade 0 (none) | 28 | 61
  Grade 1 (minimal) | 46 | 58
  Grade 2 (mild) | 51 | 14
  Grade 3 (moderate) | 10 | 1
  Grade 4 (severe) | 0 | 0

22. Other Pre Specified Outcome: Erythema
Description: as for outcome 18
Time Frame: 4 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 132
participants
  Grade 0 (none) | 54 | 72
  Grade 1 (minimal) | 54 | 49
  Grade 2 (mild) | 24 | 11
  Grade 3 (moderate) | 3 | 0
  Grade 4 (severe) | 0 | 0

23. Other Pre Specified Outcome: Erythema
Description: as for outcome 18
Time Frame: 8 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 132 | 129
participants
  Grade 0 (none) | 79 | 81
  Grade 1 (minimal) | 30 | 39
  Grade 2 (mild) | 18 | 7
  Grade 3 (moderate) | 5 | 2
  Grade 4 (severe) | 0 | 0

24. Other Pre Specified Outcome: Erythema
Description: as for outcome 18
Time Frame: 12 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 132 | 130
participants
  Grade 0 (none) | 80 | 85
  Grade 1 (minimal) | 34 | 36
  Grade 2 (mild) | 15 | 8
  Grade 3 (moderate) | 3 | 1
  Grade 4 (severe) | 0 | 0

25. Other Pre Specified Outcome: Edema
Description: EDEMA SCALE Grade 0 = None Grade 1 = Minimal - scant, rare edema Grade 2 = Mild - easily seen edema, minimally palpable, involving up to 1/3 of the treatment area Grade 3 = Moderate - easily seen edema and typically palpable, involving between 1/3 to 2/3 of the treatment area Grade 4 = Severe - easily seen edema, indurated in some areas, involving over 2/3 of the treatment area
Time Frame: Baseline
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants
  Grade 0 (none) | 133 | 134
  Grade 1 (minimal) | 2 | 0
  Grade 2 (mild) | 0 | 0
  Grade 3 (moderate) | 0 | 0
  Grade 4 (severe) | 0 | 0

26. Other Pre Specified Outcome: Edema
Description: as for outcome 25
Time Frame: 5 minutes after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants
  Grade 0 (none) | 92 | 127
  Grade 1 (minimal) | 30 | 7
  Grade 2 (mild) | 10 | 0
  Grade 3 (moderate) | 3 | 0
  Grade 4 (severe) | 0 | 0

27. Other Pre Specified Outcome: Edema
Description: as for outcome 25
Time Frame: 24-48 hours after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants
  Grade 0 (none) | 89 | 133
  Grade 1 (minimal) | 27 | 0
  Grade 2 (mild) | 18 | 1
  Grade 3 (moderate) | 1 | 0
  Grade 4 (severe) | 0 | 0

28. Other Pre Specified Outcome: Edema
Description: as for outcome 25
Time Frame: 2 weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants
  Grade 0 (none) | 131 | 134
  Grade 1 (minimal) | 4 | 0
  Grade 2 (mild) | 0 | 0
  Grade 3 (moderate) | 0 | 0
  Grade 4 (severe) | 0 | 0

29. Other Pre Specified Outcome: Edema
Description: as for outcome 25
Time Frame: 4 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 132
participants
  Grade 0 (none) | 134 | 132
  Grade 1 (minimal) | 1 | 0
  Grade 2 (mild) | 0 | 0
  Grade 3 (moderate) | 0 | 0
  Grade 4 (severe) | 0 | 0

30. Other Pre Specified Outcome: Edema
Description: as for outcome 25
Time Frame: 8 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 132 | 129
participants
  Grade 0 (none) | 131 | 128
  Grade 1 (minimal) | 0 | 0
  Grade 2 (mild) | 1 | 0
  Grade 3 (moderate) | 0 | 1
  Grade 4 (severe) | 0 | 0

31. Other Pre Specified Outcome: Edema
Description: as for outcome 25
Time Frame: 12 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 132 | 130
participants
  Grade 0 (none) | 132 | 130
  Grade 1 (minimal) | 0 | 0
  Grade 2 (mild) | 0 | 0
  Grade 3 (moderate) | 0 | 0
  Grade 4 (severe) | 0 | 0

32. Other Pre Specified Outcome: Stinging/Burning
Description: STINGING AND BURNING SCALE Grade 0 = None Grade 1 = Minimal, barely perceptible -tolerable and little discomfort Grade 2 = Moderate - tolerable, but causes some discomfort Grade 3 = Severe - very uncomfortable or intolerable
Time Frame: Baseline
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants
  Grade 0 (none) | 134 | 133
  Grade 1 (mild) | 1 | 0
  Grade 2 (moderate) | 0 | 1
  Grade 3 (severe) | 0 | 0

33. Other Pre Specified Outcome: Stinging/Burning
Description: as for outcome 32
Time Frame: During PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants
  Grade 0 (none) | 10 | 111
  Grade 1 (mild) | 39 | 23
  Grade 2 (moderate) | 74 | 0
  Grade 3 (severe) | 12 | 0

34. Other Pre Specified Outcome: Stinging/Burning
Description: as for outcome 32
Time Frame: 5 minutes after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants
  Grade 0 (none) | 30 | 130
  Grade 1 (mild) | 70 | 4
  Grade 2 (moderate) | 35 | 0
  Grade 3 (severe) | 0 | 0

35. Other Pre Specified Outcome: Stinging/Burning
Description: as for outcome 32
Time Frame: 24-48 Hours after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants
  Grade 0 (none) | 107 | 132
  Grade 1 (mild) | 23 | 2
  Grade 2 (moderate) | 5 | 0
  Grade 3 (severe) | 0 | 0

36. Other Pre Specified Outcome: Stinging/Burning
Description: as for outcome 32
Time Frame: 2 Weeks after PDT #1
Population: ITT
Measure: Number; unit: ITT
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
ITT
  Grade 0 (none) | 131 | 134
  Grade 1 (mild) | 3 | 0
  Grade 2 (moderate) | 0 | 0
  Grade 3 (severe) | 1 | 0

37. Other Pre Specified Outcome: Stinging/Burning
Description: as for outcome 32
Time Frame: 4 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 132
participants
  Grade 0 (none) | 132 | 132
  Grade 1 (mild) | 2 | 0
  Grade 2 (moderate) | 1 | 0
  Grade 3 (severe) | 0 | 0

38. Other Pre Specified Outcome: Stinging/Burning
Description: as for outcome 32
Time Frame: 8 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 132 | 129
participants
  Grade 0 (none) | 130 | 129
  Grade 1 (mild) | 2 | 0
  Grade 2 (moderate) | 0 | 0
  Grade 3 (severe) | 0 | 0

39. Other Pre Specified Outcome: Stinging/Burning
Description: as for outcome 32
Time Frame: 12 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 132 | 130
participants
  Grade 0 (none) | 130 | 130
  Grade 1 (mild) | 1 | 0
  Grade 2 (moderate) | 1 | 0
  Grade 3 (severe) | 0 | 0

40. Other Pre Specified Outcome: Scaling & Dryness
Description: SCALING AND DRYNESS SCALE Grade 0 = None Grade 1 = Minimal - barely perceptible desquamation Grade 2 = Mild - limited areas of fine desquamation in up to 1/3 of the treatment area Grade 3 = Moderate - fine desquamation involving 1/3 to 2/3 of the treatment area or limited areas of coarser scaling Grade 4 = Severe - coarser scaling involving more than 2/3 of the treatment area or limited areas of very coarse scaling
Time Frame: Baseline
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants
  Grade 0 (none) | 83 | 78
  Grade 1 (minimal) | 35 | 41
  Grade 2 (mild) | 10 | 11
  Grade 3 (moderate) | 7 | 4
  Grade 4 (severe) | 0 | 0

41. Other Pre Specified Outcome: Scaling & Dryness
Description: as for outcome 40
Time Frame: 24-48 hours after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants
  Grade 0 (none) | 84 | 79
  Grade 1 (minimal) | 30 | 40
  Grade 2 (mild) | 17 | 10
  Grade 3 (moderate) | 4 | 5
  Grade 4 (severe) | 0 | 0

42. Other Pre Specified Outcome: Scaling & Dryness
Description: as for outcome 40
Time Frame: 2 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants
  Grade 0 (none) | 33 | 81
  Grade 1 (minimal) | 47 | 38
  Grade 2 (mild) | 29 | 11
  Grade 3 (moderate) | 26 | 4
  Grade 4 (severe) | 0 | 0

43. Other Pre Specified Outcome: Scaling & Dryness
Description: as for outcome 40
Time Frame: 4 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 132
participants
  Grade 0 (none) | 73 | 83
  Grade 1 (minimal) | 44 | 38
  Grade 2 (mild) | 15 | 11
  Grade 3 (moderate) | 3 | 0
  Grade 4 (severe) | 0 | 0

44. Other Pre Specified Outcome: Scaling & Dryness
Description: as for outcome 40
Time Frame: 8 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 132 | 129
participants
  Grade 0 (none) | 83 | 86
  Grade 1 (minimal) | 35 | 35
  Grade 2 (mild) | 11 | 5
  Grade 3 (moderate) | 3 | 3
  Grade 4 (severe) | 0 | 0

45. Other Pre Specified Outcome: Scaling & Dryness
Description: as for outcome 40
Time Frame: 12 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 132 | 130
participants
  Grade 0 (none) | 85 | 86
  Grade 1 (minimal) | 33 | 32
  Grade 2 (mild) | 9 | 10
  Grade 3 (moderate) | 5 | 2
  Grade 4 (severe) | 0 | 0

46. Other Pre Specified Outcome: Oozing/Vesiculation/Crusting
Description: OOZING/VESICULATION/CRUSTING Grade 0 = None Grade 1 = Minimal - a single area of oozing, vesiculation or crusting 3 mm diameter or less in size Grade 2 = Mild - two to four areas of oozing, vesiculation or crusting 3 mm diameter or less in size OR a single area larger than 3 mm diameter in size Grade 3 = Moderate - more than a single area of oozing, vesiculation or crusting larger than 3 mm diameter in size or more than four areas of 3 mm diameter or less in size Grade 4 = Severe - any degree of oozing, vesiculation or crusting greater than (3) above
Time Frame: Baseline
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants
  Grade 0 (none) | 128 | 129
  Grade 1 (minimal) | 7 | 4
  Grade 2 (mild) | 0 | 1
  Grade 3 (moderate) | 0 | 0
  Grade 4 (severe) | 0 | 0

47. Other Pre Specified Outcome: Oozing/Vesiculation/Crusting
Description: as for outcome 46
Time Frame: 24-48 hours after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants
  Grade 0 (none) | 116 | 127
  Grade 1 (minimal) | 12 | 3
  Grade 2 (mild) | 5 | 3
  Grade 3 (moderate) | 2 | 1
  Grade 4 (severe) | 0 | 0

48. Other Pre Specified Outcome: Oozing/Vesiculation/Crusting
Description: as for outcome 46
Time Frame: 2 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 134
participants
  Grade 0 (none) | 92 | 129
  Grade 1 (minimal) | 23 | 4
  Grade 2 (mild) | 16 | 1
  Grade 3 (moderate) | 4 | 0
  Grade 4 (severe) | 0 | 0

49. Other Pre Specified Outcome: Oozing/Vesiculation/Crusting
Description: as for outcome 46
Time Frame: 4 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 135 | 132
participants
  Grade 0 (none) | 121 | 129
  Grade 1 (minimal) | 12 | 2
  Grade 2 (mild) | 2 | 1
  Grade 3 (moderate) | 0 | 0
  Grade 4 (severe) | 0 | 0

50. Other Pre Specified Outcome: Oozing/Vesiculation/Crusting
Description: as for outcome 46
Time Frame: 8 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 132 | 129
participants
  Grade 0 (none) | 125 | 124
  Grade 1 (minimal) | 5 | 3
  Grade 2 (mild) | 2 | 2
  Grade 3 (moderate) | 0 | 0
  Grade 4 (severe) | 0 | 0

51. Other Pre Specified Outcome: Oozing/Vesiculation/Crusting
Description: as for outcome 46
Time Frame: 12 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA-PDT | Vehicle
Number analyzed (Participants) | 132 | 130
participants
  Grade 0 (none) | 123 | 125
  Grade 1 (minimal) | 5 | 4
  Grade 2 (mild) | 3 | 0
  Grade 3 (moderate) | 1 | 1
  Grade 4 (severe) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | ALA-PDT | Vehicle
Serious Adverse Events (participants affected / at risk) | 5/135 | 2/134
Other Adverse Events (participants affected / at risk) | 6/135 | 6/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALA-PDT (N=135) | Vehicle (N=134)
Angina Unstable (Cardiac disorders) | 1 (1) | 0 (0)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0
Chest Pressure (Cardiac disorders) | 1 (1) | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ALA-PDT (N=135) | Vehicle (N=134)
Nasopharyngitis (Infections and infestations) | 2 | 4
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication of results from multi-center trial will be made by the Sponsor. If publication is not submitted within 12 months after conclusion of the study, the PI may publish the results from the site individually, subject to compliance with the other terms of the clinical trial agreement, including a requirement that the PI provide a draft of the publication for the sponsor's review 30-75 days before submission so that sponsor can review the publication for confidential information.